CLINICAL TRIAL: NCT07069530
Title: Impact of Musical Therapeutic Intervention on Depression in Dementia Patients and Caregiver Burden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida SouthWestern State College (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Hieu Nguyen, Principle Investigator, Florida SouthWestern State College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Music-2025; #FSWHRP2022-1-29-01 (Other: Florida SouthWestern State College Institutional Review Board)
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Dementia; Alzheimer Disease (AD); Depression Chronic; Caregiver Burden of People With Dementia; Cognitive Impairments
Keywords: Music Therapy; Dementia; Depression; Alzheimer's Disease; Caregiver Burden; Receptive Music Intervention
MeSH Terms: conditions — Dementia; Alzheimer Disease; Cognitive Dysfunction; Depression; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music Therapy Intervention Arm (Experimental): Participants in this arm received six 30-minute sessions of receptive live music therapy delivered via solo piano performance over the course of two weeks. Sessions were held in a communal setting one hour before dinner, using a fixed playlist to ensure consistency. Pre- and post-intervention measures included the Geriatric Depression Scale (GDS) for residents and the Caregiver Burden Scale in End-of-Life Care (CBS-EOLC) for staff.
  Interventions: Behavioral: Receptive Music Therapy

INTERVENTIONS:
Behavioral: Receptive Music Therapy — Participants received six 30-minute sessions of receptive music therapy delivered by live solo piano performance over two weeks. The same playlist was performed in a fixed order at each session, held one hour before dinner. The intervention was designed to reduce depressive symptoms in dementia patients and alleviate caregiver burden using a structured, low-cost, non-pharmacological approach.

SUMMARY:
This single-site interventional study evaluated the effects of receptive live music therapy on depression in patients with dementia and caregiver burden at the AMAVIDA Memory Care Unit in Fort Myers, Florida. Over two weeks, participants attended six 30-minute live piano performances using a fixed setlist delivered one hour before dinner. Pre- and post-intervention assessments included the Geriatric Depression Scale (GDS) for patients and the Caregiver Burden Scale in End-of-Life Care (CBS-EOLC) for staff caregivers. Data were analyzed using paired-sample t-tests to compare depression and burden scores before and after the music intervention.

DETAILED DESCRIPTION:
This exploratory study was designed to assess the feasibility and therapeutic potential of receptive live music as a non-pharmacological intervention for older adults with dementia and their caregivers in a residential memory care setting. The intervention involved structured, live piano performances using a fixed repertoire and delivery schedule to maintain consistency across sessions. Participants were recruited from a licensed memory care unit within a retirement community at Amavida in Fort Myers Florida and included both residents diagnosed with Alzheimer's disease or related dementias and their long-term caregivers.

Eligible residents underwent cognitive screening using the Mini-Mental State Examination (MMSE) to ensure the ability to engage meaningfully with the intervention. Pre- and post-intervention assessments focused on psychological well-being, specifically depression and caregiver burden. Validated scales-the 15-item Geriatric Depression Scale (GDS) and the Caregiver Burden Scale in End-of-Life Care (CBS-EOLC)-were administered to quantify changes in mental health outcomes.

Music sessions occurred in a communal space and were integrated into the facility's daily schedule one hour prior to dinner. Caregivers remained present but unobtrusive during performances to minimize interference. Data were collected confidentially, and participants were informed of their right to withdraw at any time.

The study emphasized ecological validity by embedding the intervention in a real-world care environment without modifying existing pharmacological treatment plans. Findings were analyzed using standard statistical methods to determine within-subject change.

ELIGIBILITY:
Inclusion Criteria:

* Resident participants must be aged 60 or older.
* Residents must have a documented diagnosis of Alzheimer's disease or related dementia.
* Residents must have completed a Mini-Mental State Examination (MMSE) with a score of ≥17.
* Caregiver participants must be aged 25 or older.
* Caregivers must have at least one year of experience working in the memory care unit.

Exclusion Criteria:

* Residents with MMSE scores <17 indicating severe cognitive impairment.
* Residents unable to provide coherent verbal responses.
* Participants (residents or caregivers) who decline to provide informed consent.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Geriatric Depression Scale (GDS) Score Among Residents | Within 2 weeks (pre- and post-intervention)
  The Geriatric Depression Scale (Short Form, 15 items) was administered to residents diagnosed with dementia before and after a two-week receptive music therapy intervention. Scores range from 0 to 15, with higher scores indicating greater depressive symptoms. The primary outcome is the change in GDS score from pre- to post-intervention.

SECONDARY OUTCOMES:
Change in Caregiver Burden Scale in End-of-Life Care (CBS-EOLC) Score | Within 2 weeks (pre- and post-intervention)
  The Caregiver Burden Scale in End-of-Life Care (CBS-EOLC) is a validated 16-item self-report questionnaire that measures physical, emotional, and logistical strain experienced by caregivers. Scores range from 16 to 64, with higher scores indicating greater perceived burden. The secondary outcome is the change in caregiver burden scores from before to after the two-week music therapy intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hieu D Nguyen, Associates Degree, Principal Investigator — Stanford University
Locations (1):
- Amavida Assisted Living, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the small sample size and the sensitive nature of the study population, which includes cognitively impaired older adults. The data collected, including EEG readings and behavioral assessments, may pose a risk of re-identification even after de-identification procedures. Furthermore, participants and/or their legal guardians did not provide consent for their data to be shared with external researchers. The study was designed for internal use only and not intended for secondary analysis or broader data dissemination.